CLINICAL TRIAL: NCT01936441
Title: Menopausal Strategies: Finding Lasting Answers for Symptoms and Health (MsFLASH) 04: A Pilot Trial of Telephone-Based Cognitive-Behavioral Therapy for Midlife Women With Menopause-related Sleep Disturbance
Brief Title: MsFLASH-04: Pilot Trial: Telephone Behavioral Therapy for Menopause-related Sleep Disturbance
Acronym: MsFLASH-04
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MsFLASH-04; 1U01AG032699-01 (NIH)
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Hot Flashes; Menopause; Vasomotor Disturbance; Sleep
Keywords: Menopause; Vasomotor; Symptoms; Sleep; Cognitive Behavioral Therapy
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy-Insomnia (CBT-I) (Experimental): Participants will have contact with a menopause counselor 6 times over 8 weeks. The first session will be in-person at a private research office. All other contacts will be by telephone. Women unable to attend the in-person session will receive a phone call. All in-person and telephone consultations will be 20-30 minutes.
  Participants will receive reading materials before each phone call relating to menopausal changes, menopausal changes in sleep and strategies for lessening menopause related sleep disturbances. A daily sleep diary will be completed each week during the 8-week intervention period. The day before each telephone session, the participant will email that week's completed diary to a secure email address accessible only by the counselor; women who are unable to use email will provide their data by telephone directly to the counselor. During the weekly telephone calls, the reading and materials will be discussed and the sleep diary will be reviewed.
  Interventions: Behavioral: Cognitive Behavioral Therapy-Insomnia (CBT-I)
- Menopause Education Control (MEC) (Placebo Comparator): Participants will have contact with a menopause counselor 6 times over 8 weeks. The first session will be in-person at a private research office. All other contacts will be by telephone. Women who are unable to attend the in-person session will receive a phone call. All in-person and telephone consultations are designed to last 20-30 minutes. Participants will receive information about menopausal changes and ways to develop symptom management strategies. Women in the MEC will keep a daily sleep diary. The day before each telephone session, the participant will email that week's completed diary to a secure email address accessible only by the counselor; women who are unable to use email will provide their data by telephone directly to the counselor. During the weekly telephone calls, the reading material will be discussed and the sleep diary will be reviewed.
  Interventions: Behavioral: Menopause Education Control (MEC)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy-Insomnia (CBT-I) — See Experimental Arm Description
  Arms: Cognitive Behavioral Therapy-Insomnia (CBT-I)
Behavioral: Menopause Education Control (MEC) — See Experimental Arm Description
  Arms: Menopause Education Control (MEC)

SUMMARY:
Self-reported sleep complaints are common in peri- and postmenopausal women and have been identified as a key symptom of the menopausal transition. The MsFLASH study, A Pilot Trial of Telephone-Based Cognitive-Behavioral Therapy for Midlife Women with Menopause-related Sleep Disturbance, is a randomized, single-blind, placebo-controlled, two arm clinical trial. The target population will include women in general good health, aged 40-65 years, who report symptoms of insomnia (trouble sleeping) and who are bothered by hot flashes. We plan to enroll 100 women from Seattle, Washington and surrounding areas into the trial. Half of the women will be randomly assigned to receive the behavioral intervention and half to receive the behavioral control.

The intervention arm participants will receive 6 sessions of a telephone-based, cognitive-behavioral therapy intervention for insomnia (CBT-I), based on state-of-the-art methods and specifically targeted to women with menopause-related sleep disturbance (CBT-I). The control arm participants will receive telephone-based Menopause Education Control (MEC) that includes elements of sleep hygiene. Assessments for both groups will be collected at baseline (pre-randomization), 8-week post-randomization, and 6-month post-randomization.

The inclusion/exclusion criteria are designed to target broadly those midlife women who have menopause-related sleep disturbance and also report being bothered by vasomotor symptoms. This target population defines the clinical population seeking treatment for relief of menopause-related sleep problems. Exclusion criteria are kept minimal and intended only to exclude women with significant medical problems likely to account for their sleep problems (instead of menopause), or likely to interfere with their ability to participate in the intervention. We include women taking hormone therapy or other medication who meet these criteria because they are part of the population seeking clinical care for relief of sleep disturbances.

Our primary objective is to develop an intervention that is generalizable to the greatest number of women and maximally translatable into real-world primary care practice.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 40-65 years old
* Postmenopausal or perimenopausal, including:

  * Women with a uterus who have skipped 2 or more menstrual cycles with an amenorrhea interval >=60 days in the past 12 months
  * Women without a uterus or who have had a bi-lateral oophorectomy
* Experiencing hot flashes
* Experiencing insomnia (trouble sleeping) that is related to menopause
* Written informed consent signed

Exclusion Criteria:

* Pregnancy, intending pregnancy, or breastfeeding
* Current use of alcohol that is greater than 3 drinks per day
* Ever diagnosed for sleep apnea, restless legs syndrome, periodic leg movement disorder, random eye movement (REM) behavior disorder, or narcolepsy by a health care provider
* A job in the past month or planning to have a job in the next 3 months that requires shift work more than 3 times a week that involves working at night or on a rotating shift schedule
* Significant current major illness interfering with sleep or intervention participation (such as active cancer)
* Use of any prescription sleep medications more than 3 times a week or prescription medications that may affect sleep
* Use of over-the-counter medications more than three times a week that are specifically for sleep, such as Tylenol PM, Nytol, Sominex, Tranquil Nighttime Sleep Aid, Unisom, ZzzQuil, benedryl, melatonin, valerian root, alcohol
* Current participation in another intervention study
* Inability or unwillingness to complete study procedures

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Insomnia Symptoms | 8 weeks
  The primary outcome is insomnia symptoms as assessed by the Insomnia Severity Index (ISI). The primary objective of this pilot trial is to determine the efficacy of Cognitive Behavioral Therapy-Insomnia (CBT-I) vs. Menopause Education Control (MEC) in improving insomnia symptoms among mid-life women with menopause-related sleep disturbance. 24-week follow-up will be additionally assessed.

SECONDARY OUTCOMES:
Sleep Quality | 8 weeks
  The secondary outcome is self-reported sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI). 24-week follow-up will be additionally assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Guthrie, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Andrea Z LaCroix, PhD, Principal Investigator — University of California, San Diego; Susan M McCurry, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Diem SJ, LaCroix AZ, Reed SD, Larson JC, Newton KM, Ensrud KE, Woods NF, Guthrie KA. Effects of pharmacologic and nonpharmacologic interventions on menopause-related quality of life: a pooled analysis of individual participant data from four MsFLASH trials. Menopause. 2020 Oct;27(10):1126-1136. doi: 10.1097/GME.0000000000001597. PMID 32701665
- [Derived] Guthrie KA, Larson JC, Ensrud KE, Anderson GL, Carpenter JS, Freeman EW, Joffe H, LaCroix AZ, Manson JE, Morin CM, Newton KM, Otte J, Reed SD, McCurry SM. Effects of Pharmacologic and Nonpharmacologic Interventions on Insomnia Symptoms and Self-reported Sleep Quality in Women With Hot Flashes: A Pooled Analysis of Individual Participant Data From Four MsFLASH Trials. Sleep. 2018 Jan 1;41(1):zsx190. doi: 10.1093/sleep/zsx190. PMID 29165623
- [Derived] McCurry SM, Guthrie KA, Morin CM, Woods NF, Landis CA, Ensrud KE, Larson JC, Joffe H, Cohen LS, Hunt JR, Newton KM, Otte JL, Reed SD, Sternfeld B, Tinker LF, LaCroix AZ. Telephone-Based Cognitive Behavioral Therapy for Insomnia in Perimenopausal and Postmenopausal Women With Vasomotor Symptoms: A MsFLASH Randomized Clinical Trial. JAMA Intern Med. 2016 Jul 1;176(7):913-20. doi: 10.1001/jamainternmed.2016.1795. PMID 27213646